CLINICAL TRIAL: NCT00547807
Title: Non-Nutritive Sucking and Swaddling for Pain Relief in Term Neonates: a Randomised Controlled Trial
Brief Title: Non-Nutritive Sucking and Swaddling for Pain Relief in Term Neonates: Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sociedade Hospital Samaritano (Other)
Responsible Party: Mariana Bueno, HCFMUSP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS 52/06
Record Dates: First submitted 2007-10-22; First posted 2007-10-23 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Pain
Keywords: Pain, neonate, nursing care
MeSH Terms: conditions — Pain | interventions — Complementary Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non-nutritive sucking — Non-nutritive sucking is applied by using a gloved finger
  Other Names: complementary therapy
Other: Swaddling — Swaddling is an age-old practice of wrapping infants snugly in swaddling cloths, blankets or similar cloth so that movement of the limbs is tightly restricted

SUMMARY:
Non pharmacological approaches are important in pain control in neonates, specially in term healthy neonates. Non-nutritive sucking and swaddling are considered effective strategies for pain control in these population, but the effect in their association are not clear until now. The hypothesis of the study is that association between non-nutritive sucking and swaddling reduces pain scores resulting from venepuncture compared to non-nutritive sucking alone.

ELIGIBILITY:
Inclusion Criteria:

* Term healthy neonates

Exclusion Criteria:

* NICU admission

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
pain score | pre painfull procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Bueno, MSN, Principal Investigator — Sociedade Hospital Samaritano; Edna A Bussotti, RN, Principal Investigator — Sociedade Hospital Samaritano; Andréia Silva, RN, Principal Investigator — Sociedade Hospital Samaritano
Locations (1):
- Sociedade Hospital Samaritano, São Paulo, São Paulo, Brazil